CLINICAL TRIAL: NCT03893526
Title: The Effect of Neprilysin on Plasma Concentrations of Glucagon-Like Peptide-1 in Patients With Type 2 Diabetes
Brief Title: Effect of Neprilysin on Glucagon-Like Peptide-1 in Patients With Type 2 Diabetes
Acronym: NEPT2D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Nicolai Jacob Wewer Albrechtsen, Resident, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEPT2D
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Type2 Diabetes
Keywords: GLP-1; Neprilysin; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — sacubitril and valsartan sodium hydrate drug combination; Sitagliptin Phosphate; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants are subjected to a standardized meal
  Interventions: Drug: Placebo
- Entrestro (Active Comparator): 194 mg sacubitril / 206 mg valstartan (entresto) as one single dose followed by a standardized meal
  Interventions: Drug: Entresto
- Sitagliptin (Active Comparator): 200mg sitagliptin (100mg the night before and 100mg on the study day) as one single dose followed by a standardized meal
  Interventions: Drug: Sitagliptin
- Entrestro + sitagliptin (Active Comparator): 194 mg sacubitril / 206 mg valstartan (entresto) + 200mg sitagliptin (100mg the night before and 100mg on the study day) as one single dose followed by a standardized meal
  Interventions: Drug: Entresto; Drug: Sitagliptin
- Valsartan (Active Comparator): 206mg valsartan as one single dose followed by a standardized meal
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Entresto — Single dose administration of entresto
  Arms: Entrestro; Entrestro + sitagliptin
Drug: Sitagliptin — Single dose administration of sitagliptin
  Arms: Entrestro + sitagliptin; Sitagliptin
Drug: Valsartan — single doses administration of valsartan
  Arms: Valsartan
Drug: Placebo — placebo day
  Arms: Placebo

SUMMARY:
Glucagon-like peptide-1(GLP-1) is secreted during a meal and increases glucose induced insulin secretion. The enzyme dipeptidyl peptidase 4(DPP-4) cleaves intact GLP-1 within minutes and DPP-4 inhibitors are therefore used for treatment of diabetic hyperglycemia. A few animal studies have implicated the enzyme neutral endopeptidase 24.11 (24.11) in the degradation of GLP-1 but if this is the case in humans with type 2 diabetes is unknown.

We therefore administered a NEP inhibitor, 194mg sacubitril, a DPP-4 inhibitor (sitagliptin 100mg the night before and 100mg 2 hours before), both, or placebo, to patients with type 2 diabetes during a standardized meal and measured plasma concentrations of GLP-1

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Oral Antidiabetics Medicine Only
* Body Mass Index of 25-35
* Type 2 Diabetes

Exclusion Criteria:

* acute diseases within the two weeks
* chronic diseases
* smoker
* alcoholism, drug addiction or recent weight loss
* blood donation within the last 3 months

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 3 hours after treatment ( during the subsequent standardized meal)
  Plasma Concentrations of glucose

SECONDARY OUTCOMES:
Plasma Concentrations of GLP-1 | 3 hours after treatment ( during the subsequent standardized meal)
Plasma Concentrations of GIP | 3 hours after treatment ( during the subsequent standardized meal)
Plasma Concentrations of Glucagon | 3 hours after treatment ( during the subsequent standardized meal)
Plasma Concentrations of Insulin | 3 hours after treatment ( during the subsequent standardized meal)
Plasma Concentrations of C-Peptide | 3 hours after treatment ( during the subsequent standardized meal)
Plasma Concentrations of Amino Acids | 3 hours after treatment ( during the subsequent standardized meal)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, RegionH, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Wewer Albrechtsen NJ, Moller A, Martinussen C, Gluud LL, Rashu EB, Richter MM, Plomgaard P, Goetze JP, Kjeldsen S, Hansen LH, Gustafsson F, Deacon CF, Holst JJ, Madsbad S, Bojsen-Moller KN. Acute effects on glucose tolerance by neprilysin inhibition in patients with type 2 diabetes. Diabetes Obes Metab. 2022 Oct;24(10):2017-2026. doi: 10.1111/dom.14789. Epub 2022 Jul 21. PMID 35676803